CLINICAL TRIAL: NCT01253525
Title: A Phase 1b Study of Weekly Paclitaxel With Ramucirumab (IMC-1121B) Drug Product in Patients With Advanced Gastric Adenocarcinomas
Brief Title: Study of Weekly Paclitaxel With Ramucirumab in Participants With Advanced Gastric Adenocarcinomas
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14204; CP12-1026 (Other: ImClone Systems); I4T-IE-JVBW (Other: Eli Lilly and Company)
Record Dates: First submitted 2010-12-02; First posted 2010-12-03 (Estimated); Results first posted 2014-06-18 (Estimated); Last update posted 2014-06-18 (Estimated); Status verified 2014-05

CONDITIONS: Adenocarcinoma
Keywords: Adenocarcinoma; Gastroesophageal Junction
MeSH Terms: conditions — Adenocarcinoma | interventions — Ramucirumab; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ramucirumab (IMC-1121B ) and Pacitaxel (Experimental): Each treatment cycle is 4 weeks (28 days)
  Interventions: Biological: Ramucirumab (IMC-1121B ); Drug: Paclitaxel

INTERVENTIONS:
Biological: Ramucirumab (IMC-1121B ) — 8 milligrams/kilogram (mg/kg) intravenously on Days 1 and 15 of each 28-ay cycle
  Other Names: LY3009806; IMC-1121B
Drug: Paclitaxel — 80 milligram/square meter (mg/m2) intravenously Days 1, 8, and 15 of each 28 day cycle

SUMMARY:
Investigate the safety and tolerability of ramucirumab (IMC-1121B) drug product (DP) in combination with paclitaxel.

ELIGIBILITY:
Inclusion Criteria:

* Has a histopathologically or cytologically confirmed diagnosis of gastric or gastroesophageal junction (GEJ) adenocarcinoma
* Has an advanced or metastatic solid gastric adenocarcinoma that has failed standard therapy
* Has resolution of all clinically significant toxic effects of prior therapy, surgery, treatment with an investigational agent or device, treatment monoclonal antibody or small molecule, and radiotherapy or chemotherapy.
* Has adequate organ function
* Eligible participants of reproductive potential (both sexes) agree to use adequate contraceptive methods (hormonal or barrier methods) during the study period and for 12 weeks after the last dose of study medication

Exclusion Criteria:

* Has undergone major surgery within 28 days prior to the study, or subcutaneous venous access device placement within 7 days prior to the study registration date
* Has elective or planned surgery to be conducted during the trial
* Has had treatment with an investigational agent or device, an antineoplastic small molecule, or antineoplastic radiotherapy or chemotherapy
* Was previously treated with a chemotherapy regimen containing nitrosoureas or mitomycin C
* Has had treatment with an antineoplastic monoclonal antibody within 8 weeks prior to the study registration date
* Has a history of deep vein thrombosis, pulmonary embolism, or any other significant thromboembolism prior to the study registration date
* Has experienced any arterial thrombotic event, including myocardial infarction, cerebrovascular accident, or transient ischemic attack, within 6 months prior to the study date
* Is receiving therapeutic anticoagulation with warfarin, low-molecular weight heparin or similar agents. (Participants receiving prophylactic, low-dose anticoagulation therapy are eligible provided that the coagulation parameters International Normalized Ratio (INR) ≤ 1.5, prothrombin time (PT) and partial thromboplastin time (PTT) or - Is receiving chronic therapy with nonsteroidal anti-inflammatory agents [Aspirin use at doses up to 325 milligrams/day (mg/day) is permitted]
* Has significant bleeding disorders, vasculitis, history of postoperative bleeding complications, hemoptysis or had a significant bleeding episode from the gastrointestinal (GI) tract within 3 months prior to the study date
* Has a history of GI perforation and/or fistulae within 6 months prior to the study date
* Has symptomatic congestive heart failure, unstable angina pectoris, or symptomatic or poorly controlled cardiac arrhythmia
* Has uncontrolled arterial hypertension despite standard medical management.
* Has a serious or nonhealing wound or peptic ulcer or bone fracture within 28 days prior to the study date
* Has a bowel obstruction, history or presence of inflammatory enteropathy or extensive intestinal resection, Crohn's disease, ulcerative colitis, or chronic diarrhea
* Has a serious illness or medical condition(s)
* Is pregnant or lactating
* Has received treatment with another investigational drug or participation in another interventional clinical trial within 28 days prior to the study date

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2010-11; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (2):
- Japan (2):
  - ImClone Investigational Site, Chiba
  - ImClone Investigational Site, Osaka

REFERENCES:
- [Derived] Ueda S, Satoh T, Gotoh M, Gao L, Doi T. A phase ib study of safety and pharmacokinetics of ramucirumab in combination with paclitaxel in patients with advanced gastric adenocarcinomas. Oncologist. 2015 May;20(5):493-4. doi: 10.1634/theoncologist.2014-0440. Epub 2015 Apr 17. PMID 25888272

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were considered completed if they either completed Cycle 1 of study drug or discontinued study drug due to a dose limiting toxicity (DLT) during Cycle 1.
Groups:
- Ramucirumab + Paclitaxel: Ramucirumab (IMC-1121B): 8 milligrams/kilogram (mg/kg) administered intravenously on Days 1 and 15 of each 28-day cycle.
  Paclitaxel: 80 milligrams/square meter (mg/m2) administered intravenously on Days 1, 8, and 15 of each 28-day cycle.
Period: Overall Study
Arm/Group | Ramucirumab + Paclitaxel
Started | 6
Received Any Quantity of Study Drug | 6
Completed | 6
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: All enrolled participants
Arm/Group | Ramucirumab + Paclitaxel
Number analyzed (Participants) | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.6 (15.50)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 6
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 6
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Japan | 6

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a Dose-Limiting Toxicity (DLT) During Cycle 1
Description: DLT based on National Cancer Institute Common Terminology Criteria for Adverse Events (NCICTCAE v4.02) in Cycle (Cy) 1 due to study drug (SD) with (w/): Grade (Gr) ≥3 neutropenia w/fever ≥38.5°C or w/bacteremia or sepsis, thrombocytopenia w/bleeding and platelet substitution, prothrombin and/or partial thromboplastin time w/no anticoagulation, hyperbilirubinemia; Gr 4: neutropenia >5 days, thrombocytopenia, Gr 4 or uncontrollable hypertension QTc>500 milliseconds (ms) or increase ≥100 ms increase in 24 hours after SD or significant arrhythmia in this period; Gr ≥3 nonhematologic toxicity (tox), excluding Gr 3 hypersensitivity, hypertension, injection-site reaction, arthralgia/myalgia, asthenia/fatigue, diarrhea w/out loperamide/nausea/vomiting w/out antiemetic and transient aminotransferase elevation. SD tox=delay >1 week in ramucirumab (RAM) dose or omission of 1 dose of RAM or 2 paclitaxel doses due to tox in Cy 1 or delay >2 weeks between Cy 1 and Cy 2 due to persistent tox.
Time Frame: Cycle 1 of 28-day cycle
Population: All enrolled participants who complete the first cycle of study drug or discontinued study drug due to a DLT during Cycle 1.
Measure: Number; unit: participants
Arm/Group | Ramucirumab + Paclitaxel
Number analyzed (Participants) | 6
participants | 0

2. Primary Outcome: Number of Participants With Adverse Events (AEs)
Description: The number of participants who experienced AEs of any grade, AEs of Grade ≥3 or AEs resulting in death that were considered to be related to ramucirumab [RAM (IMC-1121B)] or paclitaxel (PAC). A summary of serious adverse events (SAEs) and all other non-SAEs, regardless of causality, is located in the Reported Adverse Events module.
Time Frame: Up to 47 weeks post baseline
Population: All enrolled participants who received any quantity of study drug.
Measure: Number; unit: participants
Arm/Group | Ramucirumab + Paclitaxel
Number analyzed (Participants) | 6
participants
  RAM-Related AEs Any Grade | 6
  PAC-Related AEs Any Grade | 6
  RAM-Related AEs Any Grade ≥3 | 2
  PAC-Related AEs Any Grade ≥3 | 4
  RAM-Related AEs Resulting in Death | 0
  PAC-Related AEs Resulting in Death | 0

3. Primary Outcome: Number of Participants With Serious Adverse Events (SAEs)
Description: The number of participants who experienced SAEs that were considered to be related to ramucirumab [RAM (IMC-1121B)] or paclitaxel (PAC). A summary of SAEs and all other non-SAEs, regardless of causality, is located in the Reported Adverse Events module.
Time Frame: Up to 47 weeks post baseline
Population: All enrolled participants who received any quantity of study drug.
Measure: Number; unit: participants
Arm/Group | Ramucirumab + Paclitaxel
Number analyzed (Participants) | 6
participants
  RAM-Related SAEs | 2
  PAC-Related SAEs | 2

4. Secondary Outcome: Ramucirumab Maximum Serum Concentration (Cmax) for Cycle 1
Description: Cmax after a single dose of ramucirumab (IMC-1121B).
Time Frame: Cycle 1 Pre-infusion, Days 1, 2, 3, 5, 8, 12, and 15 of 28-day cycle
Population: All enrolled participants who received any quantity of study drug and had evaluable Cmax values.
Measure: Mean (Standard Deviation); unit: micrograms/milliliter (µg/mL)
Arm/Group | Ramucirumab + Paclitaxel
Number analyzed (Participants) | 6
micrograms/milliliter (µg/mL) | 176 (46.6)

5. Secondary Outcome: Serum Anti-Ramucirumab Antibody Assessment (Immunogenicity)
Description: The percentage of participants who were treatment-emergent positive for anti-ramucirumab (IMC-1121B) antibodies.
Time Frame: Cycle 1 through Cycle 5 (28-day cycles)
Population: All enrolled participants who received at least 1 dose of study drug and were analyzed for anti-ramucirumab (IMC-1121B) antibodies.
Measure: Number; unit: percentage of participants
Arm/Group | Ramucirumab + Paclitaxel
Number analyzed (Participants) | 6
percentage of participants | 0

6. Secondary Outcome: Ramucirumab Area Under the Concentration Time Curve (AUC) for Cycle 1
Description: AUC from time 0 to infinity (0-∞) after a single dose of ramucirumab (IMC-1121B).
Time Frame: Cycle 1 Pre-infusion, Days 1, 2, 3, 5, 8, 12, and 15 of 28-day cycle
Population: All enrolled participants who received any quantity of study drug and had evaluable AUC0-∞ values.
Measure: Mean (Standard Deviation); unit: micrograms*hour/milliliter (µg*h/mL)
Arm/Group | Ramucirumab + Paclitaxel
Number analyzed (Participants) | 1
micrograms*hour/milliliter (µg*h/mL) | 34100 (NA) — Standard deviation cannot be calculated with results from 1 participant.

7. Secondary Outcome: Ramucirumab Half-Life (t1/2) for Cycle 1
Description: Terminal t1/2 (the time it takes for the concentration of ramucirumab (IMC-1121B) in plasma or serum to decline by 50%) after a single dose of ramucirumab (IMC-1121B).
Time Frame: Cycle 1: Pre-infusion, Days 1, 2, 3, 5, 8, 12, and 15 of 28-day cycle
Population: All enrolled participants who received any quantity of study drug and had evaluable t1/2 values.
Measure: Median (Full Range); unit: hours (h)
Arm/Group | Ramucirumab + Paclitaxel
Number analyzed (Participants) | 4
hours (h) | 190 [138 to 225]

8. Secondary Outcome: Ramucirumab Clearance (CL) or Cycle 1
Description: CL [the volume of plasma or serum cleared of ramucirumab (IMC-1121B) per unit time] after a single dose of ramucirumab (IMC-1121B).
Time Frame: Cycle 1: Pre-infusion, Days 1, 2, 3, 5, 8, 12, and 15 of 28-day cycle
Population: All enrolled participants who received any quantity of study drug and had evaluable CL values.
Measure: Mean (Standard Deviation); unit: liters/hour (L/h)
Arm/Group | Ramucirumab + Paclitaxel
Number analyzed (Participants) | 1
liters/hour (L/h) | 0.0166 (NA) — Standard deviation cannot be calculated with results from 1 participant analyzed.

9. Secondary Outcome: Ramucirumab Steady State Volume of Distribution (Vss) for Cycle 1
Description: Vss [distribution of ramucirumab (IMC-1121B) in the body at steady state] after a single dose of ramucirumab (IMC-1121B).
Time Frame: Cycle 1: Pre-infusion, Days 1, 2, 3, 5, 8, 12, and 15 of 28-day cycle
Population: All enrolled participants who received any quantity of study drug and had evaluable Vss values.
Measure: Mean (Standard Error); unit: liters (L)
Arm/Group | Ramucirumab + Paclitaxel
Number analyzed (Participants) | 1
liters (L) | 3.27 (NA) — Standard deviation cannot be calculated with results from 1 participant analyzed.

10. Secondary Outcome: Ramucirumab Maximum Serum Concentration (Cmax) for Cycle 2
Description: Cmax after multiple doses of ramucirumab (IMC-1121B).
Time Frame: Cycle 2: Pre-infusion, Days 1, 2, 3, 5, 8, 12, and 15 of 28-day cycle
Population: All enrolled participants who received any quantity of study drug and had evaluable Cmax values.
Measure: Mean (Standard Deviation); unit: micrograms/milliliter (µg/mL)
Arm/Group | Ramucirumab + Paclitaxel
Number analyzed (Participants) | 4
micrograms/milliliter (µg/mL) | 284 (39.7)

11. Secondary Outcome: Ramucirumab Area Under the Concentration Time Curve (AUC) for Cycle 2
Description: AUC within the dosing interval (0-τ) after multiple doses of ramucirumab (IMC-1121B).
Time Frame: Cycle 2: Pre-infusion, Days 1, 2, 3, 5, 8, 12, and 15 of 28-day cycle
Population: All enrolled participants who received any quantity of study drug and had evaluable AUC 0-τ values.
Measure: Mean (Standard Deviation); unit: micrograms*hour/milliliter (µg*h/mL)
Arm/Group | Ramucirumab + Paclitaxel
Number analyzed (Participants) | 2
micrograms*hour/milliliter (µg*h/mL) | 41900 (951)

12. Secondary Outcome: Ramucirumab Half-Life (t1/2) for Cycle 2
Description: Terminal t1/2 [the time it takes for the concentration of ramucirumab (IMC-1121B) in plasma or serum to decline by 50%] after multiple doses of ramucirumab(IMC-1121B).
Time Frame: Cycle 2: Pre-infusion, Days 1, 2, 3, 5, 8, 12, and 15 of 28-day cycle
Population: All enrolled participants who received any quantity of study drug and had evaluable t1/2 values.
Measure: Median (Full Range); unit: hours (h)
Arm/Group | Ramucirumab + Paclitaxel
Number analyzed (Participants) | 1
hours (h) | 218 [218 to 218]

13. Secondary Outcome: Ramucirumab Clearance (CL) for Cycle 2
Description: CL [the volume of plasma or serum cleared of ramucirumab (IMC-1121B) per unit time] at steady state after multiple doses of ramucirumab (IMC-1121B).
Time Frame: Cycle 2: Pre-infusion, Days 1, 2, 3, 5, 8, 12, and 15 of 28-day cycle
Population: All enrolled participants who received any quantity of study drug and had evaluable CL values.
Measure: Mean (Standard Deviation); unit: liters/hour (L/h)
Arm/Group | Ramucirumab + Paclitaxel
Number analyzed (Participants) | 2
liters/hour (L/h) | 0.0136 (0.000342)

14. Secondary Outcome: Ramucirumab Steady State Volume of Distribution (Vss) for Cycle 2
Description: Vss [distribution of ramucirumab (IMC-1121B) in in the body at steady state] is not calculated for multiple doses of ramucirumab (IMC-1121B).
Time Frame: Cycle 2: Pre-infusion, Days 1, 2, 3, 5, 8, 12, and 15 of 28-day cycle
Population: Zero participants were analyzed.
Arm/Group | Ramucirumab + Paclitaxel
Number analyzed (Participants) | 0

15. Secondary Outcome: Ramucirumab Maximum Serum Concentration (Cmax) for Cycle 3
Description: Due to sparse pharmacokinetic sampling ramucirumab (IMC-1121B) Cmax could not be calculated in Cycle 3.
Time Frame: Cycle 3: Pre-infusion, Day 1 of 28-day cycle
Population: Zero participants were analyzed.
Arm/Group | Ramucirumab + Paclitaxel
Number analyzed (Participants) | 0

16. Secondary Outcome: Ramucirumab Area Under the Concentration Time Curve (AUC) for Cycle 3
Description: Due to the sparse pharmacokinetic sampling ramucirumab (IMC-1121B) AUC within the dosing interval (0-τ) could not be calculated in Cycle 3.
Time Frame: Cycle 3: Pre-infusion, Day 1 of 28-day cycle
Population: Zero participants were analyzed.
Arm/Group | Ramucirumab + Paclitaxel
Number analyzed (Participants) | 0

17. Secondary Outcome: Ramucirumab Half-Life (t 1/2) for Cycle 3
Description: Due to sparse pharmacokinetic sampling ramucirumab (IMC-1121B) t1/2 could not be calculated in Cycle 3.
Time Frame: Cycle 3: Pre-infusion, Day 1 of 28-day cycle
Population: Zero participants were analyzed.
Arm/Group | Ramucirumab + Paclitaxel
Number analyzed (Participants) | 0

18. Secondary Outcome: Ramucirumab Clearance (CL) for Cycle 3
Description: Due to sparse pharmacokinetic sampling CL could not be calculated for ramucirumab (IMC-1121B) in Cycle 3.
Time Frame: Cycle 3: Pre-infusion, Day 1 of 28-day cycle
Population: Zero participants were analyzed.
Arm/Group | Ramucirumab + Paclitaxel
Number analyzed (Participants) | 0

19. Secondary Outcome: Ramucirumab Steady State Volume of Distribution (Vss) for Cycle 3
Description: Due to sparse pharmacokinetic sampling Vss for ramucirumab (IMC-1121B) could not be calculated in Cycle 3.
Time Frame: Cycle 3: Pre-infusion, Day 1 of 28-day cycle
Population: Zero participants were analyzed.
Arm/Group | Ramucirumab + Paclitaxel
Number analyzed (Participants) | 0

20. Secondary Outcome: Ramucirumab Maximum Serum Concentration (Cmax) for Cycle 4
Description: Due to sparse pharmacokinetic sampling ramucirumab (IMC-1121B) Cmax could not be calculated in Cycle 4.
Time Frame: Cycle 4: Pre-infusion, Day 1 of 28-day cycle
Population: Zero participants were analyzed.
Arm/Group | Ramucirumab + Paclitaxel
Number analyzed (Participants) | 0

21. Secondary Outcome: Ramucirumab Area Under the Concentration Time Curve (AUC) for Cycle 4
Description: Due to sparse pharmacokinetic sampling AUC within the dosing interval (0-τ) for ramucirumab (IMC-1121B) could not be calculated in Cycle 4.
Time Frame: Cycle 4: Pre-infusion, Day 1 of 28-day cycle
Population: Zero participants were analyzed.
Arm/Group | Ramucirumab + Paclitaxel
Number analyzed (Participants) | 0

22. Secondary Outcome: Ramucirumab Half-Life (t 1/2) for Cycle 4
Description: Due to sparse pharmacokinetic sampling t1/2 for ramucirumab (IMC-1121B) could not be calculated in Cycle 4.
Time Frame: Cycle 4: Pre-infusion, Day 1 of 28-day cycle
Population: Zero participants were analyzed.
Arm/Group | Ramucirumab + Paclitaxel
Number analyzed (Participants) | 0

23. Secondary Outcome: Ramucirumab Clearance (CL) for Cycle 4
Description: Due to sparse pharmacokinetic sampling CL for ramucirumab (IMC-1121B) could not be calculated in Cycle 4.
Time Frame: Cycle 4: Pre-infusion, Day 1 of 28-day cycle
Population: Zero participants were analyzed.
Arm/Group | Ramucirumab + Paclitaxel
Number analyzed (Participants) | 0

24. Secondary Outcome: Ramucirumab Steady State Volume of Distribution (Vss) for Cycle 4
Description: Due to sparse pharmacokinetic sampling Vss for ramucirumab (IMC-1121B) could not be calculated in Cycle 4.
Time Frame: Cycle 4: Pre-infusion, Day 1 of 28-day cycle
Population: Zero participants were analyzed.
Arm/Group | Ramucirumab + Paclitaxel
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Ramucirumab + Paclitaxel
Serious Adverse Events (participants affected / at risk) | 4/6
Other Adverse Events (participants affected / at risk) | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ramucirumab + Paclitaxel (N=6)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Pneumonia (Infections and infestations) | 2 (2)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1)
Lymphangiosis carcinomatosa (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Meningism (Nervous system disorders) | 1 (7)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ramucirumab + Paclitaxel (N=6)
Anaemia (Blood and lymphatic system disorders) | 2 (5)
Leukopenia (Blood and lymphatic system disorders) | 1 (3)
Lymphopenia (Blood and lymphatic system disorders) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 4 (7)
Hearing impaired (Ear and labyrinth disorders) | 1 (1)
Retinal haemorrhage (Eye disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 2 (4)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 3 (5)
Vomiting (Gastrointestinal disorders) | 2 (5)
Face oedema (General disorders) | 1 (1)
Fatigue (General disorders) | 2 (4)
Oedema peripheral (General disorders) | 1 (2)
Pyrexia (General disorders) | 3 (6)
Hypersensitivity (Immune system disorders) | 1 (1)
Lung infection (Infections and infestations) | 1 (1)
Onychomycosis (Infections and infestations) | 1 (1)
Skin laceration (Injury, poisoning and procedural complications) | 1 (1)
Alanine aminotransferase increased (Investigations) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 2 (2)
Blood alkaline phosphatase increased (Investigations) | 1 (1)
Blood lactate dehydrogenase increased (Investigations) | 1 (1)
Blood urine present (Investigations) | 1 (1)
Neutrophil count decreased (Investigations) | 1 (2)
Platelet count decreased (Investigations) | 2 (3)
Weight decreased (Investigations) | 1 (1)
White blood cell count decreased (Investigations) | 2 (6)
Decreased appetite (Metabolism and nutrition disorders) | 3 (4)
Hyperglycaemia (Metabolism and nutrition disorders) | 2 (2)
Hyperuricaemia (Metabolism and nutrition disorders) | 1 (1)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 2 (2)
Hypophosphataemia (Metabolism and nutrition disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Headache (Nervous system disorders) | 2 (2)
Neuropathy peripheral (Nervous system disorders) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 2 (2)
Insomnia (Psychiatric disorders) | 1 (1)
Haematuria (Renal and urinary disorders) | 1 (1)
Proteinuria (Renal and urinary disorders) | 3 (4)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 5 (8)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 3 (3)
Onychoclasis (Skin and subcutaneous tissue disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 4 (6)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1)
Hot flush (Vascular disorders) | 1 (3)
Hypertension (Vascular disorders) | 2 (3)

LIMITATIONS AND CAVEATS:
Cycle 3 and beyond pharmacokinetic sampling was collected per the protocol-defined limited sampling schedule.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigators agreed to delay independently publishing or disclosing data, findings or conclusions from the study except as part of a multi-center publication. Upon study publication or if the draft publication is not produced within approximately 6 months of the final report of the study results, investigators may independently publish, subject to confidential information review/redaction by sponsor. The sponsor may request publication delay up to 90 days to seek patent protection.